CLINICAL TRIAL: NCT06603259
Title: The Galleri® Community Research Program
Status: Enrolling by invitation | Type: Observational
Sponsor: GRAIL, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: GRAIL-MA-003
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Data Collection
Keywords: observational; Galleri test; Multi-cancer early detection; data collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
GRAIL, the company that developed the Galleri test and is sponsoring this study, would like to learn more from individuals who have received the Galleri multi-cancer early detection test.

The purpose of this study is to understand how health information can be accurately collected from the medical records of individuals who have received the Galleri test in a real world setting. The collected information may include relevant medical and cancer history, diagnostic test results, including the Galleri test result. This will help GRAIL build a future larger study for individuals who have taken the Galleri test. This future study is important for understanding patient journeys after a Galleri test (including any diagnostic testing done and any diagnoses made), for improving the Galleri test, and to contribute to other research on cancer screening.

ELIGIBILITY:
Inclusion Criteria:

* Have received the Galleri test prescribed by a provider per clinical care
* Capable of giving signed and legally effective informed consent. Consent provided by a legally authorized representative is not permitted in this protocol.
* Have signed HIPAA authorization(s)* form for their medical records to be released and used for this study.

Exclusion Criteria:

* Patients are excluded from the study if the patient is a GRAIL employee or contractor.
* Patients who have received the Galleri test in a GRAIL-sponsored research setting (i.e., clinical trial) are excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Biologically male and female at birth
Study Population: up to 250 participants who have received test results following the Galleri test in the real world setting.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Quality of data retrieved from participants who have received the Galleri test | From enrollment to the the end of study (12 month study participation period), data will be retrieved and assessed for this measure.
  Data quality is measured by data completeness and accuracy of key cancer outcome data elements retrieved from medical records for confirmed cancer cases of participants who received the Galleri test.

SECONDARY OUTCOMES:
Data retrieval methods will be described. | From enrollment to the the end of study (12 month study participation period), data will be retrieved and assessed for this measure.
  Summary of data retrieval methods, abstraction methods (e.g., manual, NLP assisted, LLM) that are used to abstract each key cancer outcome data element will be described. Additionally, the availability of each key cancer outcome data element depending on the time of abstraction following a Galleri test result will also be described.
Describe the process of recruiting and consenting patients, and the retrieval of records in a narrative summary. | From enrollment to the the end of study (12 month study participation period), data will be retrieved and assessed for this measure.
  The process of recruiting and consenting patients, and the retrieval of records will be described in a narrative summary.

CONTACTS AND LOCATIONS:
Overall Officials: Mai Tran, MPA, Principal Investigator — GRAIL, Inc.
Locations (1):
- GRAIL, Menlo Park, California, United States

IPD SHARING:
Plan to Share IPD: Undecided